CLINICAL TRIAL: NCT05378607
Title: Goals for Adherence with Low-cost Incentives
Acronym: GOALS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: IDinsight (Other); Mildmay Uganda Limited (Other)
Responsible Party: Principal Investigator, Sebastian Linnemayr, Principal Investigator, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCPCC074
Record Dates: First submitted 2022-05-08; First posted 2022-05-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: ART; HIV
Keywords: HIV; Behavior change; Health behavior; Adherence; Goal setting; Behavioral economics; Incentives
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Externally assigned sub-goals (Experimental): Participants will be eligible for prize drawings every three months based on meeting externally chosen subgoals in year 1 and maintaining 90% or more adherence in Year 2 as measured using a Wisepill device. In addition, there will be a larger prize drawing conditional on showing 90% adherence at the end of year 1 and viral suppression at the end of Year 2.
  This arm will receive the intervention 'Incentivization based on gradually increasing externally chosen adherence goals ', 'Annual adherence prize drawing', 'SMS motivational messages + reminder of prize drawing', 'Year 2 re-allocation based on year 1 performance' and the intervention 'End of Year 2 viral suppression prize drawing.'
  Interventions: Behavioral: Incentivization based on gradually increasing, externally chosen adherence goals; Behavioral: End of year 1 adherence prize drawing; Behavioral: SMS motivational messages + reminder of prize drawing; Behavioral: Year 2 re-allocation based on year 1 performance; Behavioral: End of Year 2 viral suppression prize drawing
- Participatory sub-goals (Experimental): Participants will be eligible for prize drawings every three months based on meeting self-chosen subgoals in year 1 and maintaining 90% or more adherence in Year 2 as measured using a Wisepill device. In addition, there will be a larger prize drawing at the end of Years 1 and 2 that is conditional on showing 90% adherence and viral suppression, respectively.
  This arm will receive the intervention ' Incentivization based on gradually increasing self-chosen adherence goals ', 'Annual adherence prize drawing', 'SMS motivational messages + reminder of prize drawing', 'Year 2 re-allocation based on year 1 performance' and the intervention 'End of Year 2 viral suppression prize drawing.'
  Interventions: Behavioral: End of year 1 adherence prize drawing; Behavioral: SMS motivational messages + reminder of prize drawing; Behavioral: Year 2 re-allocation based on year 1 performance; Behavioral: End of Year 2 viral suppression prize drawing; Behavioral: Incentivization based on gradually increasing self-chosen adherence goals
- Fixed goal (Experimental): Participants will be eligible for prize drawings every three months based on meeting a fixed adherence goal of 90% in year 1 and maintaining this adherence level in Year 2 as measured using a Wisepill device. In addition, there will be a larger prize drawing at the end of Years 1 and 2 that is conditional on showing 90% adherence and viral suppression, respectively.
  This arm will receive the intervention ' Incentivization based on a fixed adherence goal', 'Annual adherence prize drawing', 'SMS motivational messages + reminder of prize drawing', 'Year 2 re-allocation based on year 1 performance' and the intervention 'End of Year 2 viral suppression prize drawing.'
  Interventions: Behavioral: End of year 1 adherence prize drawing; Behavioral: SMS motivational messages + reminder of prize drawing; Behavioral: Year 2 re-allocation based on year 1 performance; Behavioral: End of Year 2 viral suppression prize drawing; Behavioral: Incentivization based on a fixed adherence goal
- Control (Placebo Comparator): This arm will be provided with Mildmay's usual standard of care. Participants will not receive a prize drawing incentive based on adherence, but they will also be asked to use the Wisepill device and receive weekly motivational messages.
  This arm will receive the intervention ' SMS motivational messages '
  Interventions: Behavioral: SMS motivational messages

INTERVENTIONS:
Behavioral: Incentivization based on gradually increasing, externally chosen adherence goals — Wisepill data on adherence will be collected remotely. Every three months, participants have a chance to participate in a prize drawing for an airtime reward of 500, 5,000, or 10,000 Ugandan Shillings if adherence matches or exceeds the subgoal chosen by the study coordinator. Subgoals will gradually increase from the participant's baseline adherence up to 90%. Prize drawings can be done during regularly scheduled clinic visits if the participant has a visit corresponding to the 3-month mark or remotely via SMS text message.
  Arms: Externally assigned sub-goals
Behavioral: End of year 1 adherence prize drawing — Participants will have a chance to participate in a prize drawing at the end of year 1 with larger prize amounts of up to 20,000 Ugandan Shillings (approximately $6), where eligibility is based on reaching 90% in the three months preceding the end of year 1.
  Arms: Externally assigned sub-goals; Fixed goal; Participatory sub-goals
Behavioral: SMS motivational messages + reminder of prize drawing — Participants will receive weekly motivational messages with a reminder of their upcoming prize drawing throughout year 1 of the study.
  Arms: Externally assigned sub-goals; Fixed goal; Participatory sub-goals
Behavioral: Year 2 re-allocation based on year 1 performance — In Year 2 of the study, participants who have reached 90% by the end of year 1 will no longer be given sub-goals and instead will be eligible for prize drawings if they maintain the fixed level of 90% or higher. Those who have not reached 90% by the end of year 1 will be allocated to the intervention group that showed the highest effectiveness in year 1.
  Arms: Externally assigned sub-goals; Fixed goal; Participatory sub-goals
Behavioral: End of Year 2 viral suppression prize drawing — Participants will have a chance to participate in a prize drawing at the end of Year 2 with larger prize amounts of up to 20,000 Ugandan Shillings (approximately $6), where eligibility is based on achieving viral suppression by the end of Year 2.
  Arms: Externally assigned sub-goals; Fixed goal; Participatory sub-goals
Behavioral: Incentivization based on gradually increasing self-chosen adherence goals — Wisepill data on adherence will be collected remotely. Every three months, participants have a chance to participate in a prize drawing for an airtime reward of 500, 5,000, or 10,000 Ugandan Shillings if adherence matches or exceeds the self-chosen subgoal. While self-chosen, subgoals are subject to a minimum threshold determined by baseline adherence working towards 90% adherence. Prize drawings can be done during regularly scheduled clinic visits if the participant has a visit corresponding to the 3-month mark or remotely via SMS text message.
  Arms: Participatory sub-goals
Behavioral: Incentivization based on a fixed adherence goal — Wisepill data on adherence will be collected remotely. Every three months, participants have a chance to participate in a prize drawing for an airtime reward of 500, 5,000 or 10,000 Ugandan Shillings if adherence matches or exceeds the fixed adherence goal of 90%. Prize drawings can be done during regularly scheduled clinic visits if the participant has a visit corresponding to the 3-month mark or remotely via SMS text message.
  Arms: Fixed goal
Behavioral: SMS motivational messages — The control group will also receive weekly motivational messages but without the reminder of the upcoming prize drawing.
  Arms: Control

SUMMARY:
GOALS is a three-year randomized control trial (RCT) aimed at testing the effectiveness of three incentive designs to improve the ART adherence of those in need of adherence support. Participants in the first treatment group (T1, n=140) will be eligible for a prize drawing every three months if they reach the adherence target set for them by the study team, gradually increasing from their baseline adherence towards 90% by the end of the year. Participants in the second treatment group (T2, n=140) will be eligible if they reach the adherence target they set for themselves (subject to reaching 90% at the end of year 1 and each target being at least as high as the previous one). Participants in the third treatment group will have a fixed adherence target of 90% and will be eligible for a prize drawing every three months if this target is reached. All treatment groups will receive weekly motivational messages and a reminder of the upcoming prize drawing. The control group (T4, n=140) will receive the usual standard of care offered by the hospital and weekly motivational messages. Primary outcomes measured using Wisepill devices are mean ART adherence and the fraction of clients with adherence of 90% or more. Secondary outcomes are viral suppression, the fraction of clients with treatment interruptions of 48hrs or more, and retention in care.

DETAILED DESCRIPTION:
Low ART adherence among youth living with HIV threatens positive treatment outcomes. Increasingly incentive interventions have targeted low adherence, yet little is known about how to best structure the incentives and associated eligibility criteria. A particular concern is that for those with low baseline performance, the often relatively high, fixed eligibility thresholds may be perceived as too difficult to reach and be demotivating for the most vulnerable. Our study tests a novel incentive design that permits even those with low initial adherence to qualify for incentives aimed at increasing ART adherence by allowing participants to win prizes for smaller subgoals that build towards a higher goal. This design is based on applications of behavioral economics' Prospect Theory to the psychological literature on goal setting and motivation, which suggests that distant goals can exert a demotivating effect on the individual compared to more proximal goals.

The study is separated into two parts. Study 1 will monitor ART adherence using Wisepill devices for three months among an expected 1,049 individuals aged 15-30 years who have been on ART for three or more months and have regular access to a mobile phone. Monitoring baseline adherence will ensure that individuals being randomized to the interventions in Study 2 are indeed those in need of adherence support, i.e. have low baseline mean adherence of less than 90%.

Study 2 will randomize an expected 560 participants with low adherence from Study 1 into one of four equal-sized intervention arms. In the three treatment arms, participants will be eligible for a prize drawing to win small amounts of mobile airtime of either 500, 5,000 or 10,000 Ugandan Shillings (approximately $0.15, $1.5 and $3) if they reach the adherence goal required in the respective treatment arm. The goals will be set as follows:

1. Assigned sub-goals: the study coordinator will choose an ART adherence target for the participant based on their baseline adherence and gradually increase the target every three months, working towards 90% adherence at the end of year 1.
2. Participatory sub-goals: the participant will choose their own adherence target every three months, working towards 90% adherence at the end of year 1.
3. Fixed goal: the study participant must reach a target adherence level of 90% every three months.
4. Control group: will receive the usual standard of care offered at Mildmay. All treatment groups will receive weekly motivational messages and a reminder of their upcoming prize drawing. Weekly SMS messages will help maintain contact with study participants and enable them to become accustomed to receiving messages from the study for potential remote prize drawings. In contrast, the control group will only receive the motivational portion of the text messages (without the reminders of the possibility of winning prizes) as an attention control due to the potential beneficial effects of the messages.

Year 1 of the three-year RCT will evaluate the relative effectiveness of the three incentive approaches for improving adherence. Participants in the three treatment arms will be eligible to enter an in-person or remote prize drawing for a mobile airtime reward every three months if they meet their target adherence. In-person prize drawings will be done if the date of the drawing coincides with the participants' regularly scheduled clinic visits; otherwise, they will be done remotely. Participants will also be eligible to enter a larger prize drawing at the end of year 1 if they reach 90% adherence. Year 2 will test the relative effectiveness of the interventions for maintaining at least 90% mean adherence. Participants will be eligible for a prize drawing every three months if they maintain 90% adherence and a larger prize drawing at the end of the year if viral suppression is attained. Participants that did not reach 90% adherence by the end of year 1 will be allocated to the treatment arm that showed the highest effectiveness in year 1. Follow-up surveys will be conducted every six months after enrolment into Study 2, and prize drawing surveys will be done at every prize drawing to understand cognitive and motivational factors that the intervention may influence. Year 3 will investigate the effectiveness of the three treatment arms on long-term adherence once incentives are removed. A cost-effectiveness analysis will also be performed to help determine the intervention design's potential for sustainability and scale-up.

ELIGIBILITY:
Inclusion Criteria:

* If the participant is between 15 and 30 years of age (inclusive),
* has received ART from Mildmay for at least three months,
* exhibits Wisepill-measured adherence of under 90%,
* and has regular access to a mobile phone (at least five days per week)

Exclusion Criteria:

* If the participant is not within the age range specified above,
* has not received ART from Mildmay for at least three months,
* cannot use a Wisepill device when taking ART medication,
* cannot follow the consenting procedures
* does not have regular access to a mobile phone (at least five days per week)
* or shows Wisepill-measured adherence of over 90%

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 560 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2027-02-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Mean adherence to ART in previous 12 months | Measured at 12 months
  Wisepill devices monitor the date and time of all device openings to retrieve ART medication, allowing ART adherence to be tracked continuously on the Wisepill server. This will be coded as the number of ART doses taken / number of doses prescribed.
Mean adherence to ART in previous 12 months | Measured at 24 months
  Wisepill devices monitor the date and time of all device openings to retrieve ART medication, allowing ART adherence to be tracked continuously on the Wisepill server. This will be coded as the number of ART doses taken / number of doses prescribed.
The fraction of clients with adherence of 90% or more | Measured at 12 months
  Wisepill devices monitor the date and time of all openings of the device to retrieve ART medication allowing adherence to be tracked continuously through the Wisepill server. The fraction of clients with 90% adherence or more from the total number of clients will be monitored.
The fraction of clients with adherence of 90% or more | Measured at 24 months
  Wisepill devices monitor the date and time of all openings of the device to retrieve ART medication allowing adherence to be tracked continuously through the Wisepill server. The fraction of clients with 90% adherence or more from the total number of clients will be monitored.

SECONDARY OUTCOMES:
Fraction of clients with treatment interruptions of more than 48 hours | Measured at 12 months
  Wisepill devices monitor the date and time of all openings of the device to retrieve ART medication, allowing the fraction of clients with treatment interruptions of more than 48 hours to be tracked continuously over the Wisepill server.
Fraction of clients with treatment interruptions of more than 48 hours | Measured at 24 months
  Wisepill devices monitor the date and time of all openings of the device to retrieve ART medication, allowing the fraction of clients with treatment interruptions of more than 48 hours to be tracked continuously over the Wisepill server.
Fraction of clients with treatment interruptions of more than 48 hours | Measured at 36 months
  Wisepill devices monitor the date and time of all openings of the device to retrieve ART medication, allowing the fraction of clients with treatment interruptions of more than 48 hours to be tracked continuously over the Wisepill server.
Suppressed viral load (viral load <=200 copies/ML) | Measured at 12 months
  Viral load will be chart abstracted from clinic data. They are typically done once a year.
Suppressed viral load (viral load <=200 copies/ML) | Measured at 24 months
  Viral load will be chart abstracted from clinic data. They are typically done once a year.
Suppressed viral load (viral load <=200 copies/ML) | Measured at 36 months
  Viral load will be chart abstracted from clinic data. They are typically done once a year.
Retention in Care | Measured at 12 months
  Retention in care will be chart abstracted from clinic data. First, we will use the binary definition from the Health Resources and Services Administration HIV/AIDS Bureau, which defines retention as at least 2 clinic visits separated by 90 days in the previous 12 months. Second, we will use the more detailed measure outlined by Lee et al. (2018) to create a variable that categorizes clients as having different levels of retention in care over the previous 12 months. This goes beyond the binary definition and provides more granular information about retention. We will define a client as fully retained in care if they attended all scheduled appointments over the previous 12 months (usually 4 or 5 total appointments). We will then create three different levels of care disengagement: missed one appointment but not more than 6 months without a visit, missed 2 appointments or 6-9 months without a visit, and missed 3 or more appointments or 9-12 months without a visit.
Retention in Care | Measured at 24 months
  Retention in care will be chart abstracted from clinic data. First, we will use the binary definition from the Health Resources and Services Administration HIV/AIDS Bureau, which defines retention as at least 2 clinic visits separated by 90 days in the previous 12 months. Second, we will use the more detailed measure outlined by Lee et al. (2018) to create a variable that categorizes clients as having different levels of retention in care over the previous 12 months. This goes beyond the binary definition and provides more granular information about retention. We will define a client as fully retained in care if they attended all scheduled appointments over the previous 12 months (usually 4 or 5 total appointments). We will then create three different levels of care disengagement: missed one appointment but not more than 6 months without a visit, missed 2 appointments or 6-9 months without a visit, and missed 3 or more appointments or 9-12 months without a visit.
Retention in Care | Measured at 36 months
  Retention in care will be chart abstracted from clinic data. First, we will use the binary definition from the Health Resources and Services Administration HIV/AIDS Bureau, which defines retention as at least 2 clinic visits separated by 90 days in the previous 12 months. Second, we will use the more detailed measure outlined by Lee et al. (2018) to create a variable that categorizes clients as having different levels of retention in care over the previous 12 months. This goes beyond the binary definition and provides more granular information about retention. We will define a client as fully retained in care if they attended all scheduled appointments over the previous 12 months (usually 4 or 5 total appointments). We will then create three different levels of care disengagement: missed one appointment but not more than 6 months without a visit, missed 2 appointments or 6-9 months without a visit, and missed 3 or more appointments or 9-12 months without a visit.
Mean adherence to ART in previous 12 months | Measured at 36 months
  Wisepill devices monitor the date and time of all device openings to retrieve ART medication, allowing ART adherence to be tracked continuously on the Wisepill server. This will be coded as the number of ART doses taken / number of doses prescribed.
The fraction of clients with adherence of 90% or more | Measured at 36 months
  Wisepill devices monitor the date and time of all openings of the device to retrieve ART medication allowing adherence to be tracked continuously through the Wisepill server. The fraction of clients with 90% adherence or more from the total number of clients will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Connor, PhD, Study Director — IDinsights
Locations (1):
- Mildmay Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data resulting from the proposed research will be shared with external researchers. Once the project is finished and the primary outcome data have been published, the data from the project will be made available for public use through the NICHD Data and Specimen Hub "DASH" (https://dash.nichd.nih.gov/). Constraints imposed by human research subjects protection regulations (e.g., HIPAA Protected Health Information) and RAND's IRB will be recognized as allowed by NIH.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the project is finished and the primary outcome data have been published, the data from the project will be made available for public use through the NICHD Data and Specimen Hub "DASH" (https://dash.nichd.nih.gov/).
Access Criteria: The data from the project will be made available for public use through the NICHD Data and Specimen Hub "DASH" (https://dash.nichd.nih.gov/). Constraints imposed by human research subjects protection regulations (e.g., HIPAA Protected Health Information) and RAND's IRB will be recognized as allowed by NIH.

REFERENCES:
- [Derived] Linnemayr S, Huang HC, Wagner Z, Onkundi FK, Mukasa B, Odiit M. Goals for Adherence with Low-cost Incentives (GOALS): a protocol for a randomized controlled trial evaluating the impact of small airtime incentives on ART adherence among young people living with HIV in Kampala, Uganda. Trials. 2023 Aug 9;24(1):511. doi: 10.1186/s13063-023-07449-z. PMID 37559069